CLINICAL TRIAL: NCT01849822
Title: A Feasibility Study of the Ability of the Neural Prosthetic System to Provide Direct Brain Control of Extracorporeal Devices in Patients With Quadriplegia Due to High Spinal Cord Injury
Brief Title: Providing Brain Control of Extracorporeal Devices to Patients With Quadriplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard A. Andersen, PhD (Other)
Collaborators: University of Southern California (Other); Rancho Los Amigos National Rehabilitation Center (Other)
Responsible Party: Sponsor-Investigator, Richard A. Andersen, PhD, James G. Boswell Professor of Neuroscience, California Institute of Technology
Organization: California Institute of Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16384
Record Dates: First submitted 2013-04-25; First posted 2013-05-09 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Tetraplegia
Keywords: neural; prosthetic; brain machine interface; brain computer interface; brain control; paralysis; tetraplegia; quadriplegia; spinal cord injury
MeSH Terms: conditions — Quadriplegia; Paralysis; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neural Prosthetic System (Experimental): The Neural Prosthetic System consists of two Neuroport Arrays, which are described in detail in the intervention description. Both Neuroport Arrays are inserted into the posterior parietal cortex, an area of the brain used in reach and grasp planning. The arrays are inserted and the percutaneous pedestal is attached to the skull during a surgical procedure. Following surgical recovery the subjects will participate in study sessions 3-5 times per week in which they will learn to control an end effector by thought. They will then use the end effector to perform various reach and grasp tasks.
  Interventions: Device: Neural Prosthetic System

INTERVENTIONS:
Device: Neural Prosthetic System — The Neural Prosthetic System is primarily composed of two NeuroPort Arrays. Each array is comprised of 100 microelectrodes (1.5 mm in length) uniformly organized on a 4 mm x 4 mm silicon base that is 0.25 mm thick. Each microelectrode is insulated with Parylene-C polymer and is electrically isolated from neighboring electrodes by non-conducting glass. Each microelectrode has a platinum tip that is 100-200 microns in length and offers impedance values from 100-800 kilo-ohms. Of the 100 electrodes, 96 are wire bonded using 25 micron gold alloy insulated wires collectively sealed with a silicone elastomer. The wire bundle is potted to a printed circuit board with epoxy, the printed circuit board is inserted into the Patient Pedestal (percutaneous connector), and then the Patient Pedestal is filled with silicone elastomer. Two fine platinum reference wires are also attached to the Patient Pedestal. The Patient Pedestal is 19 mm wide at the skin interface.
  Other Names: NeuroPort Array

SUMMARY:
This research study is being done to develop a brain controlled medical device, called a brain-machine interface or BMI, that will provide people with a spinal cord injury some ability to control an external device such as a computer cursor or robotic limb by using their thoughts.

Developing a brain-machine interface (BMI) is very difficult and currently only limited technology exists in this area of neuroscience. The device in this study involves implanting very fine recording electrodes into areas of the brain that are known to create arm movement plans and provide hand grasping information. These movement and grasp plans would then normally be sent to other regions of the brain to execute the actual movements. By tying into those pathways and sending the movement plan signals to a computer instead, the investigators can translate the movement plans into actual movements by a computer cursor or robotic limb.

The device being used in this study is called the NeuroPort Array and is surgically implanted in the brain. This device and the implantation procedure are experimental which means that it has not been approved by the Food and Drug Administration (FDA). One NeuroPort Array consists of a small grid of electrodes that will be implanted in brain tissue with a small cable that runs from the electrode grid to a small hourglass-shaped pedestal. This pedestal is designed to be attached to the skull and protrude though the scalp to allow for connection with the computer equipment.

The investigators hope to learn how safe and effective the NeuroPort Array is in controlling computer generated images and real world objects, such as a robotic arm, using imagined movements of the arms and hands. To accomplish this goal, two NeuroPort Arrays will be used.

ELIGIBILITY:
Inclusion Criteria:

* High cervical spinal lesion
* Able to provide informed consent
* Able to understand and comply with instructions in English
* Able to communicate via speech
* Surgical clearance
* Life expectancy greater than 12 months
* Live within 60 miles of study location and willing to travel up to 5 days per week
* A regular caregiver to monitor the surgical site
* Psychosocial support system

Exclusion Criteria:

* Presence of memory problems
* intellectual impairment
* Psychotic illness or chronic psychiatric disorder, including major depression
* Poor visual acuity
* Pregnancy
* Active infection or unexplained fever
* scalp lesions or skin breakdown
* HIV or AIDS infection
* Active cancer or chemotherapy
* Diabetes
* Autonomic dysreflexia
* History of seizure
* Implanted hydrocephalus shunt
* Previous neurosurgical history affecting parietal lobe function
* Medical conditions contraindicating surgery and chronic implantation of a medical device
* Prior cranioplasty
* Unable to undergo MRI or anticipated need for MRI during study
* Nursing an infant or unwilling to bottle-feed infant
* Chronic oral or intravenous use of steroids or immunosuppressive therapy
* Suicidal ideation
* Drug or alcohol dependence
* Planning to become pregnant, or unwilling to use adequate birth control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-02; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Andersen, PhD, Principal Investigator — California Institute of Technology; Charles Liu, MD, PhD, Principal Investigator — University of Southern California; Christi Heck, MD, PhD, MMM, Principal Investigator — University of Southern California; Mindy Aisen, MD, Principal Investigator — Rancho Los Amigos National Rehabilitation Center
Locations (3):
- United States (3):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Southern California, Los Angeles, California
  - California Institute of Technology, Pasadena, California

REFERENCES:
- [Derived] Bashford L, Rosenthal IA, Kellis S, Bjanes D, Pejsa K, Brunton BW, Andersen RA. Neural subspaces of imagined movements in parietal cortex remain stable over several years in humans. J Neural Eng. 2024 Aug 28;21(4):046059. doi: 10.1088/1741-2552/ad6e19. PMID 39134021
- [Derived] Saif-Ur-Rehman M, Lienkamper R, Parpaley Y, Wellmer J, Liu C, Lee B, Kellis S, Andersen R, Iossifidis I, Glasmachers T, Klaes C. SpikeDeeptector: a deep-learning based method for detection of neural spiking activity. J Neural Eng. 2019 Jul 23;16(5):056003. doi: 10.1088/1741-2552/ab1e63. PMID 31042684
- See also: Related Info — http://www.vis.caltech.edu/press
- Available data/document: Publication — http://www.vis.caltech.edu/papers — "Hand Shape Representation in Parietal Reach Region". The Journal of Neuroscience.
- Available data/document: Publication — http://www.vis.caltech.edu/papers — "Decoding motor imagery from the posterior parietal cortex of a tetraplegic human." Science

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrolled subject was recruited through Rancho Los Amigos Rehabilitation Center by the study medical investigator.
Groups:
- Neural Prosthetic System: The Neural Prosthetic System consists of two Neuroport Arrays. Both Neuroport Arrays are inserted into the posterior parietal cortex, an area of the brain used in reach and grasp planning. The arrays are inserted and the percutaneous pedestal is attached to the skull during a surgical procedure. Following surgical recovery the subjects will participate in study sessions 3-5 times per week in which they will learn to control an end effector by thought. They will then use the end effector to perform various reach and grasp tasks.
Period: Overall Study
Arm/Group | Neural Prosthetic System
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1 participant
Arm/Group | Neural Prosthetic System
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
Patient Control Over the End Effector (Virtual or Physical) [Count of Participants; unit: Participants] | 1
Absence of Infection or Irritation [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Patient Control Over the End Effector (Virtual or Physical)
Description: The primary effectiveness objective of this study is to evaluate the effectiveness of the NPS in controlling virtual or physical end effectors. The driving hypotheses are that control over the physical and virtual end effectors, as measured by accuracy, will be significantly greater than the level of chance. Three methods will be used to assess the effectiveness of the extracorporeal device: standardized tests, comparison of task performance to the level of chance, and the Quality-of-Life Inventory (QOLI). In collaboration with therapists at Rancho Los Amigos National Rehabilitation Center, two commonly-used, standard tests have been selected by which the use of robotic arm will be evaluated: the Action Research Arm Test (ARAT) and the Canadian Occupational Performance Measure (COPM).
Time Frame: Six years after array implantation
Population: tetraplegic patient
Measure: Count of Participants; unit: Participants
Arm/Group | Neural Prosthetic System
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Number of Participants With Absence of Infection or Irritation
Description: The primary objective of this study is to evaluate the safety of the NPS. The driving hypotheses are that the implantation will not be associated with infection or irritation, and that the serious adverse event rate will not rise above 1%. The method of evaluation will be inspection of subject's scalp for evidence of reddening or discharge; review of new symptoms including possible fever, headache, visual or auditory changes, or change in mood or behavior; serial neurologic exams. The condition of the area will be compared with its condition on previous visits. History will be obtained regarding new symptoms. Neurologic exam will be compared to baseline neuro exam. The SAE rate will be calculated as the number of SAEs per implant days.
Time Frame: Six years after array implantation
Population: Tetraplegic patient
Measure: Count of Participants; unit: Participants
Arm/Group | Neural Prosthetic System
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 6 years
Arm/Group | Neural Prosthetic System
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2012-04-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT01849822/Prot_000.pdf
  • Statistical Analysis Plan (2012-04-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT01849822/SAP_001.pdf